CLINICAL TRIAL: NCT03427723
Title: Peripheral Intravenous Cannulation in Children With Difficult Vein Access : Randomized Study Comparing Accuvein®400 Versus Standard Care
Brief Title: Accuvein Versus Standard Care for Intravenous Cannulation Procedure in Children
Acronym: AVEn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHU-374; 2017-A02975-49 (Other: 2017-A02975-49)
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Vascular Access
Keywords: Peripheral intravenous cannulation; children; near-infrared light
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: accuvein versus standard
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): visualization and palpation
  Interventions: Other: Standard care
- Accuvein (Experimental): system uses an infrared laser beam to project the image of superficial veins to the skin
  Interventions: Device: Accuvein®400

INTERVENTIONS:
Device: Accuvein®400 — The intervention comes down to the randomization of the standard treatment versus Accuvein for peripheral intravenous cannulation
  Arms: Accuvein
Other: Standard care — The intervention comes down to the randomization of the standard treatment versus Accuvein for peripheral intravenous cannulation
  Arms: Standard care

SUMMARY:
Peripheral intravenous cannulation is one of the most common procedures performed in children admitted to hospital. It is a painful and anxiety-provoking gesture for children with possible memorization of the pain even more present for patients with chronic pathology. Nevertheless, this care is essential to administer the treatments.

The cannulation is usually set up by the observation and touching of the veins by the nurse. However, this technique is often insufficient in young children and especially infants because they have a higher thickness adipose tissue. Their veins are of small caliber, hardly visible and palpable which increases the probability of a failure of the insertion of the catheter at the first attempt.

In the literature, different techniques are mentioned to promote the visualization of veins and thus the insertion of cannulation. The AccuVein®400 (AV400) system uses an infrared laser beam to project the image of superficial veins to the skin. In adults, AV400 has been shown to improve the success rate of insertion cannulation when venous capital is precarious. The question now arises as to whether this tool could be of interest to children who are particularly difficult to assist cannulation, especially the youngest of them.

Investigator hypothesize that AV400 could bring a benefit to the placement of cannulation, in the child with a venous capital difficult to catheterize and thus increase the success of the cannulation at the first attempt.

DETAILED DESCRIPTION:
Children admitted to pediatric emergencies, pediatric day hospitals and the general pediatric ward, who are less than 3 years old and whose care requires the placement of a cannulation will be identified by the caregivers as potentially included.

The DIVA score will be carried out by the nurse who takes care of the child thanks to the dedicated form. If the child has an Emla® patch, this score will be achieved after removing the patch. The nurse that will achieve the score will be the same that will pose the intravenous cannulation. Children with an assessment score <4 will not be included in the study but will still be counted.

The nurse must perform the randomization by inquiring about the randomization week: standard method or AV400 method.

The information will be made to the parents and the information form given. The parents' consent regarding the care of their child will be collected by the same nurse.

The means of prevention of pain and distraction will be set up in box with the nurse and / or the auxiliary childcare and the parents. Peripheral intravenous cannulation will be performed by the nurse in collaboration with the auxiliary childcare.

Caregivers and parents will evaluate the care. The documents concerning the practical realization of the study will be grouped together and made available in each service in dedicated bins.

ELIGIBILITY:
Inclusion Criteria:

* Child under 3 years old (male or female) managed at the University Hospital of Clermont-Ferrand with an indication of the placement of a peripheral intravenous access,
* Represented by a person having parental authority,
* Parents or holder of parental authority capable of giving their consent to the study.

Exclusion Criteria:

* Need for urgent medical care
* Care practiced by a student nurse or pediatric nurse
* Refusal of the child or the holder of parental authority.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
successful of cannulation at first attempt | At day 1 (at the moment of peripheral intravenous cannulation)
  Percentage of children whose peripheral intravenous cannulation, at first attempt, is successful.

SECONDARY OUTCOMES:
Time required to install peripheral intravenous cannulation with AV400 and with the standard method | at day 1 (at the moment of peripheral intravenous cannulation)
  time in minute for peripheral intravenous cannulation
effectiveness of the care by the nurse and the parents thanks | at day 1 (at the moment of peripheral intravenous cannulation)
  Score regarding the effectiveness of the care by the nurse and the parents thanks to the Lickert scale 5 points (from "not convinced at all" to "very convinced")
pain assessment during insertion intravenous cannulation | at day 1 (at the moment of peripheral intravenous cannulation)
  Score regarding pain during insertion intravenous cannulation by an hetero scale of pain assessment : FLACC (Face Legs Activity Cry Consolability). Validated scale for acute pain during a care for children from 0 to 7 years
Success rate according to the cannulation installation site | at day 1 (at the moment of peripheral intravenous cannulation)
  percentage of successful of cannulation according to the cannulation installation site

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France